CLINICAL TRIAL: NCT05340244
Title: GE Cardiovascular Ultrasound Device Evaluation
Brief Title: GE CVUS Device Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 217021760
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Results first posted 2022-11-23 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Echocardiography
Keywords: Transthoracic Echocardiography; Transesophageal Echocardiography

STUDY DESIGN:
Intervention Model Description: This is a pre-market, open label, prospective, non-randomized clinical research study conducted at one site in the United States.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Arm 1: Experimental (Experimental)
  Interventions: Device: Investigational ultrasound exam

INTERVENTIONS:
Device: Investigational ultrasound exam — Eligible subjects will be enrolled into the study and positioned for their ultrasound exam. Standard clinical practice procedures will be followed using the standard of care device at the site to complete the clinically indicated exams.
  After the clinically indicated exam, portions of the TTE and/or TEE exam will be repeated with the investigational ultrasound device.

SUMMARY:
The purpose of the study is to collect user feedback on the Vivid E95 ultrasound system and probes during clinical procedures on the device's intended population in order to optimize the device.

DETAILED DESCRIPTION:
The purpose of the study is to collect user feedback on the Vivid E95 ultrasound system and probes during clinical procedures on the device's intended population in order to optimize the device. The primary objective of this study is to collect user feedback and de-identified images from the Vivid E95 ultrasound system and probes in TTE and TEE exams in a clinical setting. User feedback will include workflow, performance, user preference, image quality, device features, and open-ended feedback. The safety objective of this study is to collect safety information, including type and number of adverse events and device issues.

This is a pre-market, open label, prospective, non-randomized clinical research study conducted at one site in the United States. This study is not intended to support a comparative claim or test any hypotheses, such as superiority or non-inferiority. No clinical efficacy endpoints will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical indication for a TEE and/or TTE procedure with an ultrasound device
* Has a weight of at least 5kg
* Are able and willing to comply with study procedures
* If less than 7 years old, has a parent or legally authorized representative able and willing to provide written consent to participate
* If 7-17 years old, are able and willing to provide written assent to participate AND have a parent or legally authorized representative able and willing to provide written consent to participate
* If 18 years old or older, are able and willing to provide written consent to participate

Exclusion Criteria:

* Pregnant or suspected to be pregnant based on the opinion of a clinician investigator
* Expected to be at increased risk due to study participation (e.g. due to sensitivities, relative or absolute contraindication to TEE), in the opinion of a clinician investigator
* Previously participated in this study or are enrolled in another research study that could be expected to interfere with participation in study procedures
* History of esophageal surgery or known vascular ring

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Experimental
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1: Experimental
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of User Feedback Surveys
Description: The primary objective of this study is to collect user feedback from the investigational ultrasound system in TTE and TEE exams in a clinical setting. User Surveys consist of Likert scales and qualitative feedback and this data will not follow a statistical analysis plan.
Time Frame: The total number of User Surveys will be reported. Surveys capture feedback from the device user across multiple subjects. The protocol did not require surveys be collected at specific timepoints. The device was used on each subject for about 15 minutes.
Measure: Number; unit: Completed User Survey
Arm/Group | Arm 1: Experimental
Number analyzed (Participants) | 8
Completed User Survey | 1

2. Primary Outcome: Number of De-identified Images
Description: The primary objective of this study is to collect de-identified images from the investigational ultrasound system in TTE and TEE exams in a clinical setting.
Time Frame: The total number of images collected will be reported. Multiple images are collected from each subject and the protocol does not require images to be collected at specific points in time. The device was used on each subject for about 15 minutes.
Measure: Number; unit: Images Collected
Arm/Group | Arm 1: Experimental
Number analyzed (Participants) | 8
Images Collected | 329

3. Other Pre Specified Outcome: Number of Safety Events
Description: The number of adverse events will be reported. No clinical efficacy endpoints will be assessed.
Time Frame: The total number of adverse events will be reported. Subjects were monitored for adverse events throughout the duration (start to conclusion) of each investigational ultrasound exam, an average of 15 minutes per subject.
Measure: Number; unit: Adverse events
Arm/Group | Arm 1: Experimental
Number analyzed (Participants) | 8
Adverse events | 0

4. Other Pre Specified Outcome: Number of Device Issues
Description: The number of device issues will be reported. No clinical efficacy endpoints will be assessed.
Time Frame: The total number of device issues will be reported. Study staff monitored for device issues throughout the duration (start to conclusion) of each investigational ultrasound exam, an average of 15 minutes per subject.
Measure: Number; unit: device issues
Arm/Group | Arm 1: Experimental
Number analyzed (Participants) | 8
device issues | 0

ADVERSE EVENTS:
Time Frame: The subjects were monitored for adverse events throughout the duration (start to conclusion) of each investigational ultrasound exam, an average of 15 minutes.
Description: As per the study protocol, this study employed the Adverse Event (AE) and Serious Adverse Event (SAE) definitions of ISO14155:2020.
Arm/Group | Arm 1: Experimental
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT05340244/Prot_000.pdf